CLINICAL TRIAL: NCT06315582
Title: Surgical Approach to Uterine Septum: A Randomized Controlled Trial
Brief Title: Surgical Approach to Uterine Septum
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Northwestern University (Other)
Responsible Party: Principal Investigator, Magdy Milad, MD, Chief of Minimally Invasive Gynecologic Surgery in the Department of Obstetrics and Gynecology at Northwestern University, Northwestern University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: STU00220487
Record Dates: First submitted 2024-02-27; First posted 2024-03-18 (Actual); Last update posted 2025-04-27 (Actual); Status verified 2025-04

CONDITIONS: Uterine Septum; Surgical Complication; Septum; Uterus; Treatment Side Effects; Treatment
MeSH Terms: conditions — Septate Uterus | interventions — Electrosurgery

STUDY DESIGN:
Intervention Model Description: Randomized single blinded study
Who Masked: Participant, Care Provider
Masking Description: Participants will be randomized using www.randomizer.org algorithm. They will be assigned to arm in the operating room where they will get that intervention. When they get to Post Anesthesia Care Unit, they will be unblinded. Surgeon will be blinded until patient is in operating room and envelope with randomization is opened.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Study Intervention A (control group) (Active Comparator): Hysteroscopic septoplasty utilizing bipolar electrosurgery
  Interventions: Procedure: Hysteroscopic septoplasty utilizing bipolar electrosurgery
- Study Intervention B (study group) (Experimental): Hysteroscopic septoplasty utilizing scissors without electrosurgery followed by hysteroscopic morcellation of residual tissue
  Interventions: Procedure: Removal of uterine septum with hysteroscopic scissors without electrosurgery.

INTERVENTIONS:
Procedure: Removal of uterine septum with hysteroscopic scissors without electrosurgery. — Hysteroscopic septoplasty utilizing scissors without electrosurgery followed by hysteroscopic morcellation of residual tissue
  Arms: Study Intervention B (study group)
Procedure: Hysteroscopic septoplasty utilizing bipolar electrosurgery — Hysteroscopic septoplasty utilizing bipolar electrosurgery
  Arms: Study Intervention A (control group)

SUMMARY:
The objective of this study is to determine if the use of scissors without electrosurgery is superior to bipolar electrosurgery for resection of uterine septum. The investigators will be comparing procedure-level variables such as operative time, complications, and need for additional procedures.

DETAILED DESCRIPTION:
This study is being done to compare two different surgical techniques that can be used to remove the uterine septum. At Northwestern, both procedures are done routinely. Surgeon preference and comfort dictates which is offered. Both techniques are thought to achieve the same goal of removing the participants septum with a procedure called a hysteroscopy in which the participants are taken to the operating room and a scope with a camera is inserted inside their uterus while it is expanded with sterile water. The difference is the instrument used to remove the septum. One technique uses scissors without electricity or heat followed by removal of the excess tissue with a thin tube using suction. The other technique uses an electrical loop (electrosurgery) to cut and remove the tissue. The investigators will be comparing these two procedures by measuring things such as operative time, cost, and the amount of fluid (saline) the participants body absorbs. As mentioned above, to visualize the inside of the participants uterus, the investigators will expand it by filling it with saline.Some of this fluid is absorbed by the walls of the uterus and is routinely measured. This will be one of the measurements used to compare the two surgical techniques.

About 4 weeks after the participants procedure they will have a routine follow up visit to determine if there is any septum left. The investigators will do this by doing an in-office hysteroscopy at this appointment. This might be a simple vaginal ultrasound, ultrasound with saline or a follow up hysteroscopy. If there remains some septum, it would be removed during a second hysteroscopy. It is common to need a second or even third procedure to completely remove the septum. The investigators anticipate the two techniques being compared will have similar success rates in removing the uterine septum, although there is some data to suggest that the current standard of care procedure which is using electrosurgery could cause additional adhesive disease and require another procedure to remove the adhesions. Currently, there is little data comparing these two techniques and so this study will help us understand if one causes more adhesions or not.

ELIGIBILITY:
Inclusion criteria

* Have a confirmed septum (>1.0 cm) confirmed with 3D imaging and/or MRI
* 20-44 years old

Exclusion criteria

* Known tubal disease
* Bleeding diastasis
* No blood thinners
* No concurrent laparoscopy scheduled
* Patient with confirmed fibroids over >1 cm FIGO (International Federation of Gynecology and Obstetrics) type 1

Ages: 22 Years to 44 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Estimated)
Dates: Start 2024-03-11 (Actual); Primary Completion 2025-08-26 (Estimated); Study Completion 2026-02-26 (Estimated)

PRIMARY OUTCOMES:
Procedure-level variables: operative time hysteroscopic septoplasty | During the intervention/procedure/surgery
  We will measure time it takes to conduct procedure
Procedure-level variables: Surgical Cost | During the surgery
  We will compare amount of money spent.
Procedure-level variables: Fluid deficit | During the surgery
  We will measure amount of fluid deficit which is a number that is generate by hysteroscope.
Resolution of uterine septum | Assess at 4 weeks post-op hysteroscopy
  Compare septum resolution defined by being less than 1 cm in depth from the intertubal line and need for additional intervention following hysteroscopic septoplasty utilizing these two surgical techniques

SECONDARY OUTCOMES:
Compare adverse events | Immediate period-- 1 week post-operation
  Characterize and compare any potential adverse events related to the two surgical techniques for hysteroscopic septoplasty
Comparing patient recovery and satisfaction | 2 days postop
  Comparing patient recovery and satisfaction with follow up post-operative phone calls with standardized questions

CONTACTS AND LOCATIONS:
Locations (1):
- Northwestern Medicine Prentice Women's Hospital, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Fatehi Hassanabad A, Zarzycki AN, Jeon K, Dundas JA, Vasanthan V, Deniset JF, Fedak PWM. Prevention of Post-Operative Adhesions: A Comprehensive Review of Present and Emerging Strategies. Biomolecules. 2021 Jul 14;11(7):1027. doi: 10.3390/biom11071027. PMID 34356652
- [Background] Carrera M, Perez Millan F, Alcazar JL, Alonso L, Caballero M, Carugno J, Dominguez JA, Moratalla E. Effect of Hysteroscopic Metroplasty on Reproductive Outcomes in Women with Septate Uterus: Systematic Review and Meta-Analysis. J Minim Invasive Gynecol. 2022 Apr;29(4):465-475. doi: 10.1016/j.jmig.2021.10.001. Epub 2021 Oct 11. PMID 34648934
- [Background] LaMonica R, Pinto J, Luciano D, Lyapis A, Luciano A. Incidence of Septate Uterus in Reproductive-Aged Women With and Without Endometriosis. J Minim Invasive Gynecol. 2016 May-Jun;23(4):610-3. doi: 10.1016/j.jmig.2016.02.010. Epub 2016 Feb 23. PMID 26922877
- [Background] Kalaitzopoulos DR, Themeli MZ, Grigoriadis G, Alterio MD, Vitale SG, Angioni S, Daniilidis A. Fertility, pregnancy and perioperative outcomes after operative hysteroscopy for uterine septum: a network meta-analysis. Arch Gynecol Obstet. 2024 Mar;309(3):731-744. doi: 10.1007/s00404-023-07109-2. Epub 2023 Jun 24. PMID 37354236
- [Background] Practice Committee of the American Society for Reproductive Medicine. Electronic address: ASRM@asrm.org; Practice Committee of the American Society for Reproductive Medicine. Uterine septum: a guideline. Fertil Steril. 2016 Sep 1;106(3):530-40. doi: 10.1016/j.fertnstert.2016.05.014. Epub 2016 May 25. PMID 27235766
- [Background] Dason ES, Mathur S, Murji A. Hysteroscopic septoplasty: many techniques, little evidence. Fertil Steril. 2021 Nov;116(5):1426-1427. doi: 10.1016/j.fertnstert.2021.09.001. Epub 2021 Oct 1. No abstract available. PMID 34607705
- [Background] Budden A, Abbott JA. The Diagnosis and Surgical Approach of Uterine Septa. J Minim Invasive Gynecol. 2018 Feb;25(2):209-217. doi: 10.1016/j.jmig.2017.07.017. Epub 2017 Jul 26. PMID 28755995
- [Background] Yang L, Wang L, Chen Y, Guo X, Miao C, Zhao Y, Li L, Zhang Q. Cold scissors versus electrosurgery for hysteroscopic adhesiolysis: A meta-analysis. Medicine (Baltimore). 2021 Apr 30;100(17):e25676. doi: 10.1097/MD.0000000000025676. PMID 33907137